CLINICAL TRIAL: NCT00645489
Title: A Family Intervention for Improving Self-Care of Patients With Heart Failure
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: US Department of Veterans Affairs (U.S. Federal Agency)
Responsible Party: Sayers, Steven - Principal Investigator, Department of Veterans Affairs
Organization: VA Office of Research and Development (U.S. Federal Agency)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: MIRECC002; 01008; 0008
Record Dates: First submitted 2008-03-24; First posted 2008-03-27 (Estimated); Last update posted 2010-01-06 (Estimated); Status verified 2008-12

CONDITIONS: Heart Failure, Congestive
Keywords: heart failure intervention
MeSH Terms: conditions — Heart Failure | interventions — Waiting Lists

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Other): Control condition is wait-list control.
  Interventions: Other: wait list
- 2 (Experimental): Active treatment condition: psychoeducational intervention for patients with HF
  Interventions: Behavioral: psychoeducational

INTERVENTIONS:
Behavioral: psychoeducational — Psychoeducation intervention includes information about self-care of heart failure, and a communication training intervention for patients and family members
  Arms: 2
Other: wait list — Wait list
  Arms: 1

SUMMARY:
This is a pilot study of a family-based educational program for patients with heart failure, and their family members.

DETAILED DESCRIPTION:
1. Objectives(s): We plan to conduct a feasibility pilot trial of the Family Partnership Intervention (FPI) compared to patients in the HF Wait-list (WL) condition. We plan to demonstrate feasibility, estimate variances of major outcome variables, and to obtain preliminary estimates of effect sizes in preparation for subsequent grant applications. We will be able to develop a cost-effectiveness model for the relative benefit of FPI vs. no family-based for use in longer-term studies.
2. Research Design: This is a short-term, randomized clinical trial which will involve assessments for participants in the FPI condition at a pre-intervention Baseline point, immediately post-intervention, and 6 months post-intervention. Participants in the WL condition will be assessed at Baseline, undergo an approximately 8 week waiting period, and then the FPI. A longer follow-up is not planned based on the purpose of this study as a feasibility trial.
3. Methodology: We plan to randomize 40 Veterans and their family members to either the FPI condition or WL condition, in equal proportions. We will recruit patients with at least Stage C Heart Failure (NYHA class I - IV) from the Cardiology clinic of the Philadelphia VAMC. FPI will involve 4-6 hours of intervention delivered over a period of 6-8 weeks. Assessments at a pre-treatment baseline point, 8 weeks (immediately post-treatment), and 6 months will cover the following domains: a) patients' demographic characteristics and clinical functioning, b) self-care, including self-management of symptoms, knowledge of HF, and adherence to medication and dietary intake of sodium, c) measures of family functioning relevant to the medical care of the patient, and d) health care utilization costs. Primary outcome measures will be patients' self-reported HF self-care and health care utilization costs. We anticipate that patients in the FPI condition will exhibit better self-care over time compared to patients in the WL condition. We also anticipate that patients and family members will exhibit an improved family environment and better HF knowledge.

ELIGIBILITY:
Inclusion Criteria:

1. Stage C Heart Failure,[34] which refers to past or current symptoms of heart failure with underlying structural heart disease. Indicated by chronic systolic dysfunction (left ventricle [LV] ejection fraction < 45%), diastolic dysfunction (with echo evidence of diminished compliance of the LV), or both.
2. The patient's cardiologist has recommended or initiated one of the following to prevent decompensation: continuing diuretic treatment, fluid restrictions, and/or restriction/reduction of dietary sodium intake.
3. A family member or members available for study participation with whom patient lives for at least 5 days a week. Emphasis will be given to the closest family members available (i.e., spouse).
4. Subjects are able to give informed consent (see below for exclusion due to well-documented dementia or evidence of cognitive impairment).
5. Patients will be age 50 or above. Younger patients may have a different family environment than the most common type of patient who is the target of the FPI intervention.

Exclusion Criteria:

1. Patient has a well-documented diagnosis of dementia
2. Moderate or greater cognitive impairment, based on the Blessed Test of Orientation, Memory, and Concentration (BOMC)[26] score of 16.
3. Patient's family member has BOMC score of 10 (i.e., mild or greater cognitive impairment).
4. Inability to communicate verbally, major visual impairment, uncorrected hearing loss.
5. Patient and/or family member reports "frequent use" illicit substance abuse within the past year. Scores on the AUDIT-C 4 indicating alcohol abuse/dependence.[30]
6. Patient or family member has a current diagnosis of schizophrenia spectrum psychiatric disorder (e.g., schizophrenia, schizoaffective disorder).
7. Patient indicates active suicidal ideation and evaluated as a clinical risk.
8. Patient is in the Philadelphia VAMC home-telehealth program or some other incompatible intervention.
9. Patient has an unstable medical condition that would likely prevent the subject from completing the study.

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2008-03; Primary Completion 2009-03 (Actual); Study Completion 2009-12 (Actual)

PRIMARY OUTCOMES:
dietary sodium intake | 6 months

SECONDARY OUTCOMES:
medication adherence | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Steven L. Sayers, PhD, Principal Investigator — VA Medical Center, Philadelphia
Locations (1):
- VA Medical Center, Philadelphia, Philadelphia, Pennsylvania, United States